CLINICAL TRIAL: NCT00623142
Title: The Effects of Hyperbaric Oxygen Preconditioning On Cardiovascular Protection & Ischemic Reperfusion Injury
Brief Title: The Protective Effects Of Treatment With Hyperbaric Oxygen Prior To Bypass Heart Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: North of England Medical & Hyperbaric Services (Unknown)
Responsible Party: Dr. Jeysen Zivan Yogaratnam, Hull & East Yorkshire NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R0047; 04/Q1104/26
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Myocardial Reperfusion Injury; Cytoprotection
Keywords: Myocardial protection; Ischemic Reperfusion Injury; Hyperbaric Oxygen; Preconditioning
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Patients in this arm were not treated with HBO prior to CABG
- B (Experimental): Patients in this arm were treated with HBO prior to CABG
  Interventions: Drug: Hyperbaric Oxygen

INTERVENTIONS:
Drug: Hyperbaric Oxygen — 100% Oxygen at 2.4 ATA for 30 minutes followed by 5 minutes break followed by 100% Oxygen at 2.4 ATA for another 30 minutes. This intervention was given about 4 to 5 hours prior to CABG
  Other Names: Hyperbaric Oxygen Preconditioning
  Arms: B

SUMMARY:
The purpose of this study was to determine if treating patients who have coronary heart disease with hyperbaric oxygen (HBO) prior to coronary artery bypass graft (CABG) surgery reduces injury to the heart and vascular system during and after surgery. Furthermore, this study also aims to identify some of the post CABG clinical effects of HBO treatment prior to CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective first time CABG
* Patients with at least 1 vessel coronary artery disease undergoing on- pump CABG

Exclusion Criteria:

* Age ≤ 20 years or ≥ 85 years
* Ejection fraction < 30%
* Unstable angina
* Recent myocardial infarction (< 1 month)
* Any additional cardiac disease (e.g. arrythmia, aneurysm, valvular/septal disease, dissection or elevated pulmonary artery pressure)
* Any end stage organ failure (e.g. renal and respiratory failure)
* History of chronic obstructive pulmonary disease (COPD)
* Pneumothorax
* Pulmonary bullae
* Convulsions
* Current history of malignancy
* Severe myopia or intraocular lens
* Patients on K+(ATP) Channel Openers e.g. Nicorandil, Oral Hypoglycemics, Opioid Analgesics, Catecholamines.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Myocardial Hsp72 protein | Intra-operative (During CABG)
Myocardial eNOS protein | Intra-Operative (During CABG)
Serum Troponin-T | Peri-operative
Serum soluble ICAM-1 | Peri-operative
Serum soluble PSGL-1 | Peri-operative
Serum soluble P-Selectin | Peri-operative
Serum soluble E-Selectin | Peri-operative

SECONDARY OUTCOMES:
All cardiovascular haemodynamic parameters as measured by a pulmonary artery catheter | Peri-operative
Duration of mechanical ventilation | Post Operative
Duration of endotracheal intubation | post operative
Length of stay in ICU | Post-operative
Blood loss | Post operative
Inotrope usage | Post operative
Atrial Fibrillation | Post operative
Low cardiac output status | Post operative
Pulmonary complications | Post operative
Renal Complications | Post operative
Cerebrovascular complications | Post operative
Gastrointestinal complications | Post operative
Wound complications | Post operative
Cost of ICU stay | Post operative

CONTACTS AND LOCATIONS:
Overall Officials: Jeysen Z Yogaratnam, MB.BCh, BAO, MRCS, Principal Investigator — Hull & East Yorkshire NHS Trust (Castle Hill Hospital), United Kingdom
Locations (1):
- Hull & East Yorkshire NHS Trust (Castle Hill Hospital), Hull, East Riding Of Yorkshire, United Kingdom

REFERENCES:
- [Background] Yogaratnam JZ, Laden G, Guvendik L, Cowen M, Cale A, Griffin S. Pharmacological preconditioning with hyperbaric oxygen: can this therapy attenuate myocardial ischemic reperfusion injury and induce myocardial protection via nitric oxide? J Surg Res. 2008 Sep;149(1):155-64. doi: 10.1016/j.jss.2007.09.003. Epub 2007 Oct 11. PMID 17996900
- [Background] Yogaratnam JZ, Laden G, Guvendik L, Cowen M, Cale A, Griffin S. Can hyperbaric oxygen be used as adjunctive heart failure therapy through the induction of endogenous heat shock proteins? Adv Ther. 2007 Jan-Feb;24(1):106-18. doi: 10.1007/BF02849998. PMID 17526467
- [Background] Yogaratnam JZ, Laden G, Madden LA, Seymour AM, Guvendik L, Cowen M, Greenman J, Cale A, Griffin S. Hyperbaric oxygen: a new drug in myocardial revascularization and protection? Cardiovasc Revasc Med. 2006 Jul-Sep;7(3):146-54. doi: 10.1016/j.carrev.2006.04.006. PMID 16945821
- [Background] Jeysen ZY, Gerard L, Levant G, Cowen M, Cale A, Griffin S. Research report: the effects of hyperbaric oxygen preconditioning on myocardial biomarkers of cardioprotection in patients having coronary artery bypass graft surgery. Undersea Hyperb Med. 2011 May-Jun;38(3):175-85. PMID 21721351
- [Derived] Yogaratnam JZ, Laden G, Guvendik L, Cowen M, Cale A, Griffin S. Hyperbaric oxygen preconditioning improves myocardial function, reduces length of intensive care stay, and limits complications post coronary artery bypass graft surgery. Cardiovasc Revasc Med. 2010 Jan-Mar;11(1):8-19. doi: 10.1016/j.carrev.2009.03.004. PMID 20129356
- See also: publication link - Abstract — https://www.ncbi.nlm.nih.gov/pubmed/?term=The+Effects+of+Hyperbaric+Oxygen+Preconditioning+On+Cardiovascular+Protection+%26+Ischemic+Reperfusion+Injury